CLINICAL TRIAL: NCT05857449
Title: To Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LPM3480392 Injection at Different Rates in Healthy Subjects in a Phase I Clinical Trial
Brief Title: An Exploratory Study of LPM3480392 at Different Infusion Rates in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: LY03014/CT-CHN-102
Record Dates: First submitted 2021-12-06; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (Experimental): Each subject receive the same dose(X1mg) of LPM3480392 in 15minutes in the first cycle, 5 minutes in the second cycle, and 2 minutes in the third cycle .
  Interventions: Drug: LPM3480392
- Part B (Experimental): Each subject receive LPM3480392 X2mg in the first cycle and LPM3480392 X3mg in the second cycle .
  Interventions: Drug: LPM3480392

INTERVENTIONS:
Drug: LPM3480392 — Intravenous infusion

SUMMARY:
This study evaluated the safety, tolerability and PK/PD characteristics of LPM3480392 injection by intravenous infusion at different rates in healthy subjects.The experiment was divided into Part A and Part B.

Part A is a open label ,three cycle , fixed sequence dosing study .Twelve healthy male subjects were planned to be enrolled, and the same dose (X1mg)of LPM3480392 injection was intravenously injected at different infusion times in different drug administration cycles.

Part B is an open label ,two cycle , fixed sequence dosing study .Ten healthy male subjects (subjects not enrolled in Part A) were given LPM3480392 injection in 2 minutes , each subject was given X2mg at the first cycle and X3mg at the second cycle .

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily signs the informed consent.
* Healthy male, aged 18-45 years (including boundary values);
* Body mass index (BMI) 19-26kg/m2 (including boundary value), weight ≥50kg;
* Subjects are willing to take contraceptive measures and promise not to donate sperm during the study period and within 90 days after administration;
* Willing to accept cold pain test, and the non-dominant hand can be soaked in ice water bath at 2℃ (± 0.3℃) for > 10s, < 120s;

Exclusion Criteria:

* Known history of allergy to any component of the investigational product or similar drugs, or allergic constitution [subjects with previous allergy to two or more foods or drugs];
* Past or present with any clinically significant disease or chronic disease of the respiratory system, circulatory system, digestive system, urinary system, reproductive system, nervous system, endocrine system, immune system, hematology, psychiatry, dermatology, orthostatic hypotension, etc.; or any disease that may interfere with the test results or interpretation of the results;
* Patients with Raynaud's syndrome;
* The skin wounds or skin diseases that may affect the cold pain test results; Sitting systolic blood pressure (SBP) < 90 mmHg, ≥ 140 mmHg or diastolic blood pressure (DBP) < 60 mmHg, ≥ 90 mmHg; subjects with heart rate < 60 beats/min, > 100 beats/min;
* QTc > 450 ms on electrocardiogram;
* Positive urine nicotine test;
* History of alcohol abuse within 3 months prior to Screening, defined as consumption of more than 14 units of alcohol per week (1 unit = 360 mL of beer, or 45 mL of spirits of 40% alcohol content, or 150 mL of wine), or a positive breath alcohol result;
* History of substance abuse or drug abuse or positive result of urine drug screening;
* Those who consume more than 100 g of xanthine-rich foods such as chocolate per day on average; those who consume more than 100 g of foods containing grapefruit and/or pomelo; those who consume more than 1000 mL of strong tea, coffee, cola and beverages containing caffeine and/or grapefruit ingredients;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Incidents of AE (including SAE) | from baseline to day7 of second or third cycle(each cycle is 4 days)
  including abnormal value of Vital signs,physical examination,laboratory tests,12-lead ECG
DEQ scores | from baseline to day2 of second or third cycle(each cycle is 4 days)
  Drug effect questionnaire
OWS scores | from baseline to day7 of second or third cycle(each cycle is 4 days)
  Opiate Withdrawal Scale

SECONDARY OUTCOMES:
AUC0-t | baseline and within 24 hours after administration
  Pharmacokinetic index
AUC0-∞ | baseline and within 24 hours after administration
  Pharmacokinetic index
Cmax | baseline and within 24hours after administration
  Pharmacokinetic index
Tmax | baseline and within 24 hours after administration
  Pharmacokinetic index
T1/2 | baseline and within 24 hours after administration
  Pharmacokinetic index
CL | baseline and within24 hours after administration
  Pharmacokinetic index
Vd | baseline and within 24 hours after administration
  Pharmacokinetic index
MRT | baseline and within 24 hours after administration
  Pharmacokinetic index
λz | baseline and within 24 hours after administration
  Pharmacokinetic index
Cold Pain Test | baseline and within 8 hours after administration
  Pharmacodynamic index
Pupillometry | baseline and within 8 hours after administration
  Pharmacodynamic index

CONTACTS AND LOCATIONS:
Locations (1):
- The second affiliated hosipital zhejiang university school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No